CLINICAL TRIAL: NCT04161131
Title: A Pilot of ONBOARD: OvercomiNg Barriers & Obstacles to Adopting Diabetes Devices for Adults With T1D
Brief Title: Overcoming Barriers and Obstacles to Adopting Diabetes Devices
Acronym: ONBOARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molly Tanenbaum (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Molly Tanenbaum, Instructor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47667; K23DK119470 (NIH); P30DK116074 (NIH)
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Results first posted 2021-06-08 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ONBOARD Intervention (Experimental): ONBOARD consists of four 60-minute sessions over 3 months. Each session will target a key barrier to CGM use: physical, data, social, and trust. Sessions will be delivered individually to participants by a doctoral level psychologist with diabetes expertise. Each session will include relevant first-person digital stories told adults to with T1D, recounting how they managed relevant CGM barriers.
  Interventions: Behavioral: ONBOARD

INTERVENTIONS:
Behavioral: ONBOARD — Session 1: Overview; Overcoming Physical Barriers (experiential wear) Session 2: Managing CGM data (cognitive restructuring) Session 3: Social barriers (problem solving) Session 4: Trust in CGM (motivational interviewing, review of prior sessions)

SUMMARY:
This study will create a comprehensive, multicomponent behavioral intervention package (ONBOARD; OvercomiNg Barriers & Obstacles to Adopting Diabetes Devices). ONBOARD will provide adults with type 1 diabetes (T1D) the skills to maximize benefit and minimize daily interference from barriers associated with continuous glucose monitoring (CGM) and increase readiness for closed loop.

DETAILED DESCRIPTION:
The proposed research will create and refine the ONBOARD intervention for CGM use. Participants will be tracked using metrics of A1c, time in glucose target range, number of days using CGM, blood glucose (BG) downloads, diabetes problem solving, diabetes distress, and technology attitudes. The investigators will examine whether ONBOARD leads to improved diabetes and psychosocial outcomes and sustained CGM use. At the end of this study, the investigators will have created and refined a comprehensive, multicomponent intervention package to promote increased and sustained uptake of CGM and increase readiness for closed loop adoption.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 18-50 years at time of screening
2. Subject is within first year of continuous glucose monitor use OR has not been using CGM regularly in the past 6 months
3. Subject has a clinical diagnosis of type 1 diabetes
4. Subject comprehends spoken and written English

Exclusion Criteria:

1. Subject has a medical disorder that in the judgment of the investigator will interfere with completion of any aspect of the protocol.
2. Subject has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Tanenbaum, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tanenbaum ML, Ngo J, Hanes SJ, Basina M, Buckingham BA, Hessler D, Maahs DM, Mulvaney S, Hood KK. ONBOARD: A Feasibility Study of a Telehealth-Based Continuous Glucose Monitoring Adoption Intervention for Adults with Type 1 Diabetes. Diabetes Technol Ther. 2021 Dec;23(12):818-827. doi: 10.1089/dia.2021.0198. PMID 34270351
- [Result] Tanenbaum ML, Messer LH, Wu CA, Basina M, Buckingham BA, Hessler D, Mulvaney SA, Maahs DM, Hood KK. Help when you need it: Perspectives of adults with T1D on the support and training they would have wanted when starting CGM. Diabetes Res Clin Pract. 2021 Oct;180:109048. doi: 10.1016/j.diabres.2021.109048. Epub 2021 Sep 14. PMID 34534592

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Stanford Research Database, at the Stanford Endocrinology Clinic, and through online type 1 diabetes social media platforms. 81 participants were screened for eligibility.
  Participation was online. Once the participants provided their consent they were prompted to complete baseline surveys and then scheduled to receive the four intervention sessions.
Groups:
- ONBOARD Intervention: ONBOARD consists of four 60-minute sessions over 3 months. Each session will target a key barrier to Continuous Glucose Monitor (CGM) use: physical, data, social, and trust. Sessions will be delivered individually to participants by a doctoral level psychologist with diabetes expertise. Each session will include relevant first-person digital stories told adults to with T1D, recounting how they managed relevant CGM barriers.
  ONBOARD: Session 1: Overview; Overcoming Physical Barriers (experiential wear) Session 2: Managing CGM data (cognitive restructuring) Session 3: Social barriers (problem solving) Session 4: Trust in CGM (motivational interviewing, review of prior sessions)
Period: Overall Study
Arm/Group | ONBOARD Intervention
Started | 28
Completed Baseline Surveys | 27
Received Intervention | 22
Completed | 22
Not Completed | 6
Not completed — Ineligible | 2
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed the baseline survey and met all eligibility criteria
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.48 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Marital Status [Count of Participants; unit: Participants]
  Single | 11
  Married | 9
  Separated | 1
  Living with someone | 5
Education [Count of Participants; unit: Participants]
  Some College | 6
  College graduate | 11
  Graduate degree | 9
Annual Family Income [Count of Participants; unit: Participants]
  <$25,000 | 3
  $25,000-50,000 | 2
  $51,000 - 75,000 | 5
  $76,000 - 100,000 | 4
  $101,000 - 125,000 | 5
  $126,000 -150,000 | 1
  $151,000 -175,000 | 3
  >$175,000 | 2
  Unknown/Declined to state | 1
Currently Using Insulin (%) [Count of Participants; unit: Participants]
  Yes | 20
  No | 6
Length of insulin pump use [Count of Participants; unit: Participants] — Population: Only 20 participants in the study are insulin pump users
  Participants
    number analyzed (Participants) | 20
    <0.5 year | 3
    0.5-<1 year | 1
    1-<2 years | 0
    2-<5 years | 1
    >5 years | 15
Pump Brand [Count of Participants; unit: Participants] — Population: Only 20 participants in the study are insulin pump users
  Participants
    number analyzed (Participants) | 20
    Medtronic | 9
    Tandem | 7
    Insulet | 4
Currently using CGM [Count of Participants; unit: Participants]
  Yes | 23
  No | 3
Length of CGM use [Count of Participants; unit: Participants] — Population: Only 23 participants in the study were using a CGM at baseline
  Participants
    number analyzed (Participants) | 23
    <0.5 years | 10
    0.5-1 year | 10
    1-2 years | 1
    >5 years | 2
CGM brand [Count of Participants; unit: Participants] — Population: Only 23 participants in the study were using a CGM at baseline
  Participants
    number analyzed (Participants) | 23
    Dexcom | 19
    Medtronic | 1
    Abbott (Freestyle) | 3
Chronic conditions other than diabetes [Count of Participants; unit: Participants] — Participants were ask if they had any other condition(s) (yes/no) besides type 1 diabetes
  Participants
    Yes | 9
    No | 17
Frequency of CGM use in the past month (per participant) [Number; unit: participants] — Population: Only 23 participants in the study were using a CGM at baseline
  participants
    1 day: number analyzed (Participants) | 23
    1 day | 1
    5 days: number analyzed (Participants) | 23
    5 days | 1
    14 days: number analyzed (Participants) | 23
    14 days | 1
    15 days: number analyzed (Participants) | 23
    15 days | 1
    19 days: number analyzed (Participants) | 23
    19 days | 1
    21 days: number analyzed (Participants) | 23
    21 days | 2
    25 days: number analyzed (Participants) | 23
    25 days | 1
    29 days: number analyzed (Participants) | 23
    29 days | 1
    30 days: number analyzed (Participants) | 23
    30 days | 14

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c)
Description: Glycated haemoglobin (HbA1c)
Time Frame: baseline, month 3
Population: Participants with measurement at baseline and month 3 are included in the analysis
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 10
percentage of HbA1c
  baseline | 7.27 (2.18)
  month 3 | 6.73 (2)

2. Secondary Outcome: Number of Participants Who Withdraw or Are Lost to Followup Over the Course of the Study
Description: The number of participants who withdraw or are lost to followup over the course of the study is used as a measure of attrition
Time Frame: Duration of study participation (up to three months)
Measure: Count of Participants; unit: Participants
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 28
Participants | 6

3. Secondary Outcome: Number of Eligible Individuals Who Agree to Participate in the Study
Description: Number of eligible individuals who agree to participate in the study out of all those approached during recruitment
Time Frame: During screening visit (up to 50 minutes)
Population: 81 individuals were assessed for eligibility
Measure: Count of Participants; unit: Participants
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 81
Participants | 28

4. Secondary Outcome: Satisfaction With Intervention Survey
Description: Participant-rated Satisfaction Survey: Individual question scores are presented, each was measured on a Likert scale (0-4), higher scores mean more satisfaction.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  Q1. Overall, how helpful was the ONBOARD program for you? | 2.95 (0.84)
  Q2.Overall, how satisfied were you with the ONBOARD program? | 3.5 (0.86)
  Q3.Overall, how satisfied were you with receiving the ONBOARD program online? | 3.55 (0.86)
  Q4. I would recommend the ONBOARD program | 3.5 (0.51)
  Q5. Overall, how satisfied were you with the number of sessions? | 3.32 (0.72)
  Q6. Overall, how satisfied were you with the length of the sessions? | 3.32 (0.89)

5. Secondary Outcome: Percentage of Time in Range of Continuous Glucose Monitor Values Between 70 and 180 mg/dL
Description: Baseline and 3-month followup continuous glucose monitor values for percent time spent between 70-180mg/dl
Time Frame: two weeks prior to starting intervention and two weeks after the intervention (average approximately 3 months)
Population: 19 participants had CGM data available for both measurements
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 19
percentage of time in range
  Pre-intervention | 71.4 (19.4)
  Post-intervention | 75.1 (20)

6. Secondary Outcome: Diabetes Distress Scale for Type 1 Diabetes
Description: Unabbreviated Scale Title: Diabetes Distress Scale for Type 1 Diabetes (T1-DDS) is a 28-item self-report scale that highlights seven critical dimensions of distress: powerlessness, management distress, hypoglycemia distress, negative social perceptions, eating distress, physician distress, and friends/family distress. A total score is calculated using the mean of all item scores. Subscale scores are calculated using the means of specific items for each subscale.
  Min Value: 1 Max Value: 6 Higher scores mean worse outcome/more distress
Time Frame: baseline, month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | 2.27 (.66)
  month 3 | 2.02 (.60)

7. Secondary Outcome: Glucose Monitoring System Satisfaction Survey (GMSS-T1D)
Description: Scale title "Glucose Monitoring System Satisfaction Survey - Type 1 Diabetes" Min:1 Max:5 Higher mean scores mean worse outcome
Time Frame: baseline, month 3
Population: Participants who completed the protocol and with data for the respective timepoints are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 21
score on a scale
  baseline | 3.88 (.56)
  month 3 | 3.93 (.44)

8. Secondary Outcome: Percentage of CGM Data Downloaded and Available for Analysis
Description: Baseline and 3-month follow-up percentage of continuous glucose monitoring values using data available from device for use in analyses.
Time Frame: two weeks prior to starting intervention and two weeks after the intervention (average approximately 3 months)
Population: 19 participants provided CGM data for both measurements
Measure: Mean (Standard Deviation); unit: percentage of CGM wear data available
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 19
percentage of CGM wear data available
  Pre-Intervention | 76.4 (29.6)
  Post-Intervention | 81.3 (23.4)

9. Secondary Outcome: Mean Glucose Level
Description: Mean glucose level from continuous glucose monitoring data at baseline and month 3
Time Frame: baseline, month 3
Population: 20 participants provided mean glucose values at baseline and month 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 20
mg/dL
  Baseline | 149.04 (33.02)
  month 3 | 147.03 (35.26)

10. Secondary Outcome: Barriers to Diabetes Device Use Survey
Description: Title: Barriers to Diabetes Device Use is a 19-item list of barriers to diabetes device use. Participants can select between 0 and 19 barriers. Examples of barriers are: cost, insurance, lack of family support, lack of support from the diabetes care team, and not liking devices on the body.
  Min: 0 Max: 19 higher scores mean a worse outcome
Time Frame: baseline, month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | 5.45 (2.28)
  month 3 | 5.5 (2.58)

11. Secondary Outcome: Diabetes Technology Attitudes Survey
Description: Title: Diabetes Technology Attitudes Survey, a 6-item survey that asks about general attitudes about the role diabetes technology in one's life and the extent to which someone finds technology helpful for managing diabetes.
  Min: 1 Max: 5 Mean Score, higher score means better outcome
Time Frame: Baseline, Month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | 3.97 (.3)
  month 3 | 4.23 (.61)

12. Secondary Outcome: Fear of Hypoglycemia - Worry Survey
Description: Scale Title: Hypoglycemia Fear Survey II - Worry Subscale is an 18-item subscale that presents a list of concerns people with diabetes sometimes have about low blood sugar. Respondents answer based on their level of worry about each item for the past 6 months. A total score is calculated by summing individual item scores.
  Min: 0 Max: 4 Higher score indicates worse outcome
Time Frame: baseline, month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | .87 (.47)
  month 3 | .89 (.49)

13. Secondary Outcome: Hypoglycemia Confidence Scale
Description: Title: Hypoglycemia Confidence Scale is a 9-item scale that asks about how confident the respondent is in managing problems with hypoglycemia in a range of situations. A total score is calculated using the mean of all item scores.
  Min: 1 Max: 4 Higher score means better outcome/more confidence
Time Frame: baseline, month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | 3.43 (.47)
  month 3 | 3.44 (.51)

14. Secondary Outcome: Technology Use For Diabetes Problem Solving Scale
Description: Scale: Technology Use For Diabetes Problem Solving Scale is a 9-item scale that asks participants to rate how often they use different types of technology (eg phone, websites, looking at graphs of their glucose data) in managing their diabetes, solving problems and finding answers to questions that arise in managing diabetes. A total score is calculated by summing all items.
  Min: 0 Max: 5 Higher score means a better outcome
Time Frame: baseline, month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | 2.36 (.71)
  month 3 | 2.35 (.8)

15. Secondary Outcome: INSPIRE Survey
Description: Title: INsulin Dosing Systems: Perceptions, Ideas, Reflections, and Expectations (INSPIRE) is a 31-item survey that assesses perceived benefits and burdens of automated insulin delivery systems. A total score is calculated by obtaining a mean score across items, then multiplying the mean score by 25 to scale total INSPIRE measure scores from 0 to 100.
  Min: 1 Max: 5 High score means more positive outcome
Time Frame: baseline, month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 22
score on a scale
  baseline | 1.96 (.66)
  month 3 | 1.92 (.68)

16. Secondary Outcome: Frequency of Blood Glucose Monitoring
Description: Frequency will be measured as the number of times a day the participant checks blood glucose level using glucose meter
Time Frame: 3 months
Population: Data were not collected for this outcome measure
Arm/Group | ONBOARD Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 months
Arm/Group | ONBOARD Intervention
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONBOARD Intervention (N=28)
diabetic ketoacidosis (DKA) (Endocrine disorders) | 1
Ascites (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT04161131/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT04161131/SAP_001.pdf
  • Informed Consent Form (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04161131/ICF_002.pdf